CLINICAL TRIAL: NCT02173184
Title: Phase III, Randomized, Double Blind, Parallel Groups, Placebo Controlled Clinical Study to Evaluate the Efficacy and Safety of the Lactobacillus Vaccine Gynevac, in the Treatment of Bacterial Vaginosis
Brief Title: Safety and Efficacy Study of Gynevac Lactobacillus Vaccine in the Treatment of Bacterial Vaginosis
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Amvac Kft. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: LATVAC 1-2013-HU
Record Dates: First submitted 2014-06-23; First posted 2014-06-24 (Estimated); Last update posted 2014-10-29 (Estimated); Status verified 2014-10

CONDITIONS: Bacterial Vaginosis
Keywords: bacterial vaginosis; Gynevac Lactobacillus vaccine
MeSH Terms: conditions — Vaginosis, Bacterial

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo vehicle (0.9% NaCl solution)
  Interventions: Biological: Placebo
- Gynevac (Experimental): Gynevac suspension for injection, a vaccine containing Lactobacillus strains 15, 34, 79, 84, 127 inactivated by formaldehyde in 0.9% NaCl solution
  Interventions: Biological: Gynevac

INTERVENTIONS:
Biological: Gynevac — 1 IM injection of Gynevac per week, for 4 weeks (five injections in total). Vaccination can take place in no less than 7 days intervals (+3 days).
  Arms: Gynevac
Biological: Placebo — 1 IM injection of Placebo per week, for 4 weeks (five injections in total). Vaccination can take place in no less than 7 days intervals (+3 days).
  Arms: Placebo

SUMMARY:
To investigate the efficacy (therapeutic response) of Gynevac vaccination following a 5-shot treatment period in patients with bacterial vaginosis, based on the Nugent Score and the Amsel criteria

ELIGIBILITY:
Inclusion Criteria:

* Adult premenopausal females, 18 years and older.
* Mentally competent patients that can comply with the study protocol and are able to complete and keep or study related material (patient diaries, etc.).
* Signed and dated written informed consent.
* Clinical diagnosis of BV according to Amsel criteria
* Gram stains Nugent Score ≥7 or Nugent Score 4-6 with the presence of clue cells
* Patient does not need an anti-infective treatment which would be required for specific treatment of vaginosis or to prevent the development of acute vaginitis and which may affect treatment outcome of BV.
* Negative pregnancy test at screening.

Exclusion Criteria:

* Patients with other infectious causes of vulvovaginitis (e.g. Vaginal candidiasis, Trichomonas vaginalis).
* Patients with another vaginal or vulvar condition, which would confound the interpretation of clinical and or therapeutic response.
* Patients who received antifungal or antimicrobial therapy (systemic or intravaginal), as part of standard clinical practice, or clinical trial, within 14 days of randomization.
* Patients who are diagnosed with a chronic inflammatory disease (Rheumatoid Arthritis, psoriasis, Crohn's disease, Coeliac disease, spondyloarthritis rheumatica etc.)
* Women who are scheduled to be under treatment during the study period for cervical intraepithelial neoplasia (CIN) or cervical carcinoma.
* Pregnancy or lactation.
* Patients with known hypersensitivity to formaldehyde.
* Patients undergoing antibiotic treatment.
* Patients with acute polyarthritis, known serious cardiac, liver, kidney diseases or unstable diabetes mellitus.
* Known abnormalities of the blood circulation or of the haemopoietic system.
* Use of any investigational drug within 30 days from randomization.
* Patients who do not abstain from use of intravaginal products for at least 7 days prior to study randomization (e.g. douches, female deodorant sprays, spermicides, condoms, tampons, and diaphragms). Patients should also refrain from using intravaginal products 3 days prior to each study visit.
* Patients who do not abstain from vaginal intercourse during at least 3 days prior to each study visit.

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 240 (Estimated)
Dates: Start 2014-06; Primary Completion 2015-04 (Estimated); Study Completion 2015-07 (Estimated)

PRIMARY OUTCOMES:
Therapeutic response | 3 weeks from the time of last vaccine administration (+3 days maximum)
  The percentage of patients with remission according to Amsel's criteria at week 7: resolution of the clinical findings assessed at baseline, and remission according to Gram stain Nugent score: score < 4 or 4 to 6 with no presence of clue cells at week 7.

SECONDARY OUTCOMES:
Clearance of BV infection according to Amsel criteria | 3 weeks from the time of last vaccine administration (+3 days maximum)
  The percentage of patients with clearance of infection according to Amsel criteria response (three of four from: physiological discharge, negative Whiff test, negative saline wet mount for clue cells and pH<4.7) in Gynevac® or placebo, at week 7.
Clearance of BV infection according to Nugent Score | 3 weeks from the time of last vaccine administration (+3 days maximum)
  The percentage of patients with clearance of infection according to Nugent Score (NS <4 or 4-6 with no presence of clue cells) in Gynevac® or placebo, at week 7.
Overall therapeutic failure | 3 weeks from the time of last vaccine administration (+3 days maximum)
  Percentage of patients whose overall therapeutic outcome is failure, defined as Amsel = cure and Nugent score ≥4 with the presence of clue cells and Amsel = failure regardless of Nugent Score, week 7.
Change in Nugent Score | 3 weeks from the time of last vaccine administration (+3 days maximum)
  Median difference between Gynevac or placebo of the change in Nugent Score from baseline to week 7.
Change in pre- and post-vaccination IgA, IL17, and IFNγ | 3 weeks from the time of last vaccine administration (+3 days maximum)
  Median difference from baseline of IgA, IL17 and IFNγ in PBMCs isolated on week 7 by participants treated with Gynevac or Placebo

OTHER OUTCOMES:
Number of participants with AEs | 3 weeks from the time of last vaccine administration (+3 days maximum)
  Number of patients with AEs by treatment group and overall. The incidence of AEs will be summarized by system organ class, severity, type of AE, relation of study drug and outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Attila Török, MD, Principal Investigator — Pannon Reprodukciós intézet
Locations (8):
- Hungary (8):
  - Kaali Institute, Budapest
  - Zsebok Zoltan Outpatient Center, Dept. of Gynecology, Budapest
  - Kaali Institute, Debrecen
  - Kaali Institute, Győr
  - Kaali Institute, Kaposvár
  - Kaali Institute, Miskolc
  - Donatella 99 Bt., Szentes
  - Pannon Reproduction Institute, Tapolca